CLINICAL TRIAL: NCT04471727
Title: A Phase 1/2 Open-label, Multicenter, Dose Escalation and Dose Expansion Study of the Safety, Tolerability, and Pharmacokinetics of HPN328 Monotherapy and HPN328 With Atezolizumab or Ifinatamab Deruxtecan (I-DXd) in Patients With Advanced Cancers Associated With Expression of Delta-like Canonical Notch Ligand 3 (DLL3).
Brief Title: A Study in Participants With Advanced Cancers Associated With Expression of DLL3 (MK-6070-001/HPN328-4001)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Harpoon Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPN328-4001; MK-6070-001 (Other: MSD ID); HPN328-4001 (Other: Harpoon Therapeutics Inc. ID)
Record Dates: First submitted 2020-07-06; First posted 2020-07-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Small-Cell Lung Cancer; Neuroendocrine Carcinoma
Keywords: Lung Cancer; Small-Cell Lung Cancer; DLL3; Harpoon; TriTAC; Prostate Cancer; Neuroendocrine Tumors; High Grade Neuroendrocrine Features; Delta Like Canonical Notch Ligand 3; T-cell Engager
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine; Lung Neoplasms; Prostatic Neoplasms; Neuroendocrine Tumors | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Gocatamig monotherapy dose escalation with 1 week dosing interval (Experimental): Participants will receive gocatamig once weekly (Q1W) via intravenous (IV) infusion during each 21-day cycle. Dose escalation may continue until one or more RDEs are identified, participant discontinuation or the Sponsor decides to stop enrollment.
  Interventions: Biological: Gocatamig
- Gocatamig monotherapy dose escalation with 2 week dosing interval (Experimental): Participants will receive gocatamig via IV infusion once every 2 weeks (Q2W) of a 28-day cycle. Dose escalation may continue until one or more RDEs are identified, participant discontinuation, or the Sponsor decides to stop enrollment.
  Interventions: Biological: Gocatamig
- Gocatamig monotherapy dose escalation with 3 week dosing interval (Experimental): Participants will receive gocatamig via IV infusion once every 3 weeks (Q3W) of a 21-day cycle. Dose escalation may continue until one or more RDEs are identified, participant discontinuation, or the Sponsor decides to stop enrollment.
  Interventions: Biological: Gocatamig
- Gocatamig dose escalation with atezolizumab (Experimental): Small cell lung cancer (SCLC) participants will receive gocatamig via IV infusion Q2W during each 28-day cycle and Atezolizumab via IV infusion every 4 weeks (Q4W) on Day 1 of each 28-day cycle. Dose escalation may continue until one or more RDEs are identified, participant discontinuation, or the Sponsor decides to stop enrollment.
  Interventions: Biological: Gocatamig; Biological: Atezolizumab
- Gocatamig dose escalation in combination with I-DXd (Experimental): SCLC participants will receive gocatamig via IV infusion Q2W during each 42-day cycle and I-DXd via IV infusion Q3W on Day 1 and Day 22 of each 42-day cycle. Dose escalation may continue until one or more RDEs are identified, participant discontinuation, or the Sponsor decides to stop enrollment.
  Interventions: Biological: Gocatamig; Biological: Ifinatamab Deruxtecan (I-DXd)

INTERVENTIONS:
Biological: Gocatamig — IV infusion
  Other Names: HPN328; MK-6070
Biological: Atezolizumab — IV infusion
  Arms: Gocatamig dose escalation with atezolizumab
Biological: Ifinatamab Deruxtecan (I-DXd) — IV infusion
  Other Names: DS-7300a; MK-2400
  Arms: Gocatamig dose escalation in combination with I-DXd

SUMMARY:
This study will investigate the maximum tolerated dose, the recommended dose for expansion (RDE), safety, efficacy, and pharmacokinetics of gocatamig alone, gocatamig with Atezolizumab and gocatamig with I-DXd in participants with advanced cancers associated with expression of Delta-like Canonical Notch Ligand 3 (DLL3).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a histologically or cytologically confirmed malignancy associated with expression of Delta-like Canonical Notch Ligand 3 (DLL3)
* Has small cell lung cancer (SCLC) which is relapsed/refractory following at least 1 prior line of systemic therapy that included platinum-based chemotherapy
* Has Neuroendocrine Prostate Cancer (NEPC; de novo or treatment-emergent) which is relapsed/refractory to standard systemic therapy
* Has high-grade neuroendocrine tumor types other than SCLC and NEPC, with at least one of the following:

  * Disease that is relapsed/refractory to standard systemic therapy
  * Disease for which standard therapy does not exist
  * Disease for which standard therapy is not considered appropriate by the Investigator
* Must be able to provide archival tissue sample or fresh biopsy tissue sample

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has untreated central nervous system (CNS) metastases
* Has a glioma or other primary CNS malignancy
* Has spinal cord compression or symptomatic/uncontrolled epidural disease
* Has a history of intracranial hemorrhage or spinal cord hemorrhage
* Has active neurologic paraneoplastic syndrome
* Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (e.g., biweekly or more frequently)
* Has active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis
* Is ongoing treatment with immunosuppressive medications (including, but not limited to, systemic corticosteroids [prednisone dose >10mg per day or equivalent], cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] alpha agents) within 2 weeks prior to initiation of treatment, or anticipation of need for systemic immunosuppressive medication during study treatment (except protocol-required pre-medications)
* Has a history of clinically significant cardiovascular disease such as myocardial infarction, symptomatic congestive heart failure (New York Heart Association > class II), and/or uncontrolled cardiac arrhythmia within 6 months of the first dose of study drug
* Has a history of arterial thrombosis (e.g., stroke or transient ischemic attack) within 6 months
* Has active viral hepatitis, defined as hepatitis A (hepatitis A virus immunoglobulin M [IgM] positive), hepatitis B (hepatitis B virus surface antigen [HbsAg] positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). HCV with undetectable virus after treatment are eligible. Hepatitis B virus (HBV) with undetectable viral load by quantitative polymerase chain reaction (PCR) are eligible.
* Has uncontrolled infection with Human Immunodeficiency Virus (HIV)-1 or HIV-2. Well-controlled HIV are eligible.
* Has a history of allogeneic stem cell transplant or solid-organ transplant
* Has had treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Has a history of severe anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Has a history of interstitial lung disease, idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT). History of radiation pneumonitis in the radiation field is permitted
* Has had treatment with other investigational drug within 3 weeks of scheduled dosing (or 5 half-lives of drug, whichever is shorter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2027-11-03 (Estimated); Study Completion 2027-11-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who experience an adverse event | Up to ~4 years
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. AEs will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTACAE) version 5.0 (American Society for Transplant and Cellular Therapy (ASTCT) grading criteria for cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS)). The percentage of participants who experience an AE in the study will be presented.
Percentage of participants who discontinue due to an adverse event | Up to ~4 years
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. AEs will be graded according to NCI CTACAE version 5.0 (ASTCT grading criteria for CRS and ICANS). The percentage of participants who discontinue due to an AE in the study will be presented.
Number of participants with dose limiting toxicity (DLT) following treatment with HPN328 as monotherapy or in combination with atezolizumab or I-DXd | Up to ~4 years
  A DLT is defined as an AE that represents a clinically significant shift from baseline and must be considered related or suspected to be related to study drug (gocatamig and/or atezolizumab or I-DXd) by the Investigator or Sponsor. AEs will be graded according to NCI CTACAE version 5.0 (ASTCT grading criteria for CRS and ICANS). The number of participants with a DLT will be presented.
Maximum concentration (Cmax) of Gocatamig | At designated time points up to ~4 years
  Cmax is the maximum concentration of the drug observed in serum. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of gocatamig.
Cmax of Atezolizumab | At designated time points up to ~4 years
  Cmax is the maximum concentration of the drug observed in serum. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of Atezolizumab.
Cmax of I-DXd | At designated time points up to ~4 years
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of I-DXd.
Time to maximum concentration (Tmax) of Gocatamig | At designated time points up to ~4 years
  Tmax is the amount of time that a drug is present at the maximum concentration observed in serum. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax of gocatamig.
Tmax of atezolizumab | At designated time points up to ~4 years
  Tmax is the amount of time that a drug is present at the maximum concentration observed in serum. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax of atezolizumab.
Tmax of I-DXd | At designated time points up to ~4 years
  Tmax is the amount of time that a drug is present at the maximum concentration observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax of I-DXd.
Area under the concentration-time curve over the dosing interval t (AUCt) of Gocatamig | At designated time points up to ~4 years
  AUC is a measure of serum drug concentration and time and is estimated as the area under the plot of serum concentration against time after drug administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine t (AUCt) of gocatamig.
AUCt of atezolizumab | At designated time points up to ~4 years
  AUC is a measure of serum drug concentration and time and is estimated as the area under the plot of serum concentration against time after drug administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine t (AUCt) of atezolizumab.
AUCt of I-DXd | At designated time points up to ~4 years
  AUC is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine t (AUCt) of I-DXd.
Area under the concentration-time curve extrapolated to infinity (AUCinf) of Gocatamig | At designated time points up to ~4 years
  AUCinf is a measure of serum drug concentration and time to infinity and is estimated as the area under the plot of serum concentration against time to infinity after drug administration. Blood samples collected at multiple timepoints post-dose will be used to determine the AUCinf of gocatamig.
AUCinf of atezolizumab | At designated time points up to ~4 years
  AUCinf is a measure of serum drug concentration and time to infinity and is estimated as the area under the plot of serum concentration against time to infinity after drug administration. Blood samples collected at multiple timepoints post-dose will be used to determine the AUCinf of atezolizumab.
AUCinf of I-DXd | At designated time points up to ~4 years
  AUCinf is a measure of plasma drug concentration and time to infinity and is estimated as the area under the plot of plasma concentration against time to infinity after drug administration. Blood samples collected at multiple timepoints post-dose will be used to determine the AUCinf of I-DXd.
Terminal half-life (t1/2) of Gocatamig | At designated time points up to ~4 years
  t1/2 is a measure of how long it takes to clear 50% of the drug from serum after reaching Cmax. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the t1/2 of gocatamig.
t1/2 of atezolizumab | At designated time points up to ~4 years
  t1/2 is a measure of how long it takes to clear 50% of the drug from serum after reaching Cmax. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the t1/2 of atezolizumab.
t1/2 of I-DXd | At designated time points up to ~4 years
  t1/2 is a measure of how long it takes to clear 50% of the drug from plasma after reaching Cmax. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the t1/2 of I-DXd.
Single dose clearance (CL) of Gocatamig | At designated time points up to ~4 years
  CL is the apparent total clearance of the drug from serum after oral administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine CL of gocatamig.
CL of atezolizumab | At designated time points up to ~4 years
  CL is the apparent total clearance of the drug from serum after oral administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine CL of atezolizumab.
CL of I-DXd | At designated time points up to ~4 years
  CL is the apparent total clearance of the drug from plasma after oral administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine CL of I-DXd.
Steady state maximum concentration (Cmax,ss) of Gocatamig | At designated time points up to ~4 years
  Cmax,ss is the maximum concentration of the drug in serum observed in serum under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax,ss of gocatamig.
Cmax,ss of atezolizumab | At designated time points up to ~4 years
  Cmax,ss is the maximum concentration of the drug observed in serum under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Css,max of atezolizumab.
Cmax,ss of I-DXd | At designated time points up to ~4 years
  Cmax,ss is the maximum concentration of the drug observed in plasma under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax,ss of I-DXd.
Steady state Ctrough (Ctrough,ss) of Gocatamig | At designated time points up to ~4 years
  Ctrough,ss is the lowest concentration reached by a drug in serum under steady state conditions before the next dose is administered. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Ctrough,ss of gocatamig.
Ctrough,ss of atezolizumab | At designated time points up to ~4 years
  Ctrough,ss is the lowest concentration reached by a drug in serum under steady state conditions before the next dose is administered. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Ctrough,ss of atezolizumab.
Ctrough,ss of I-DXd | At designated time points up to ~4 years
  Ctrough,ss is the lowest concentration reached by a drug in plasma under steady state conditions before the next dose is administered. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Ctrough,ss of I-DXd.
Steady state time to maximum concentration (Tmax,ss) of Gocatamig | At designated time points up to ~4 years
  Tmax,ss is the amount of time that a drug is present at the maximum concentration observed in serum under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax,ss of gocatamig.
Tmax,ss of atezolizumab | At designated time points up to ~4 years
  Tmax,ss is the amount of time that a drug is present at the maximum concentration observed in serum under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax,ss of atezolizumab.
Tmax,ss of I-DXd | At designated time points up to ~4 years
  Tmax,ss is the amount of time that a drug is present at the maximum concentration observed in plasma under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax,ss of I-DXd.
Area under the steady state concentration-time curve over dosing interval t (AUCt,ss) of Gocatamig | At designated time points up to ~4 years
  AUCt,ss is a measure of serum drug concentration and time and is estimated as the area under the plot of serum concentration against time after drug administration under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AUCt,ss of gocatamig.
AUCt,ss of atezolizumab | At designated time points up to ~4 years
  AUCt,ss is a measure of serum drug concentration and time and is estimated as the area under the plot of serum concentration against time after drug administration under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AUCt,ss of atezolizumab.
AUCt,ss of I-DXd | At designated time points up to ~4 years
  AUCt,ss is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AUCt,ss of I-DXd.
Steady state t1/2 (t1/2,ss) of Gocatamig | At designated time points up to ~4 years
  t1/2,ss is a measure of how long it takes to clear 50% of the drug in serum after reaching Cmax under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the t1/2,ss of gocatamig.
t1/2,ss of Gocatamig with atezolizumab | At designated time points up to ~4 years
  t1/2,ss is a measure of how long it takes to clear 50% of the drug after reaching Cmax under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the t1/2,ss of atezolizumab.
t1/2,ss of IDXd | At designated time points up to ~4 years
  t1/2,ss is a measure of how long it takes to clear 50% of the drug in plasma after reaching Cmax under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the t1/2,ss of I-DXd.
Steady state CL (CL,ss) of Gocatamig | At designated time points up to ~4 years
  CL,ss is the apparent total clearance of the drug from serum after administration under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine CL,ss of gocatamig.
CL,ss of Gocatamig with atezolizumab | At designated time points up to ~4 years
  CL,ss is the apparent total clearance of the drug from serum after administration under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine CL,ss of atezolizumab.
CL,ss of I-DXd | At designated time points up to ~4 years
  CL,ss is the apparent total clearance of the drug from plasma after administration under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine CL,ss of I-DXd.
Steady state volume of distribution (V,ss) of Gocatamig | At designated time points up to ~4 years
  V,ss is defined as the volume of distribution in serum under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the V,ss of gocatamig.
V,ss of atezolizumab | At designated time points up to ~4 years
  V,ss is defined as the volume of distribution in serum under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the V,ss of atezolizumab.
V,ss of I-DXd | At designated time points up to ~4 years
  V,ss is defined as the volume of distribution in plasma under steady state conditions. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the V,ss of I-DXd.
Steady state accumulation ratio (AC) of Gocatamig | At designated time points up to ~4 years
  AC is the ratio of accumulation of a drug in serum under steady state conditions after repeated administration as compared to a single dose. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AC of gocatamig.
AC of atezolizumab | At designated time points up to ~4 years
  AC is the ratio of accumulation of a drug in serum under steady state conditions after repeated administration as compared to a single dose. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AC of atezolizumab.
AC of I-DXd | At designated time points up to ~4 years
  AC is the ratio of accumulation of a drug in plasma under steady state conditions after repeated administration as compared to a single dose. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AC of I-DXd.

SECONDARY OUTCOMES:
Objective response rate (ORR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) (Prostate cancer clinical trials working group 3 (PCWG3) for participants with neuroendocrine prostate cancer (NEPC)) | Up to ~4 years
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. Participants with NEPC will be evaluated using PCWG3-modified RECIST v1.1. ORR will be presented.
Extra-cranial objective response rate (EC-ORR) based on modified RECIST v1.1 | Up to ~4 years
  EC-ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 considering extra-cranial disease (i.e. exclusive of brain metastases). Participants with NEPC will be evaluated using PCWG3-modified RECIST v1.1 considering extra-cranial disease. EC-ORR will be presented.
Best Overall Response (BOR) | Up to ~4 years
  BOR is defined as the participants' best disease response during the study given a hierarchy of objective response results CR: disappearance of all target lesions per RECIST 1.1 > PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1 > stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study > progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. > not all evaluated/non-PD (NE): persistence of one or more non-target lesions and/or (if applicable) maintenance of tumor marker level above the normal limits. Percentage of participants in each BOR category will be presented.
Progression-free survival (PFS) | Up to ~4 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Participants with NEPC will be evaluated using PCWG3-modified RECIST v1.1 PFS will be presented.
Extra-cranial progression free survival (EC-PFS) | Up to ~4 years
  EC-PFS is defined as the time from randomization to the first documented extra-cranial progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Participants with NEPC will be evaluated using PCWG3-modified RECIST v1.1. EC-PFS will be presented.
Overall survival (OS) | Up to ~4 years
  OS is defined as the time from first dose of study drug to death due to any cause (summarized descriptively using Kaplan Meier method). OS will be presented.
Duration of response (DOR) | Up to ~4 years
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. Participants with NEPC will be evaluated using PCWG3-modified RECIST v1.1. DOR will be presented.
Duration of extra-cranial response (EC-DOR) | Up to ~4 years
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1), EC-DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1 considering only extra-cranial disease (i.e., exclusive of brain metastases), PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. Participants with NEPC will be evaluated using PCWG3-modified RECIST v1.1. EC-DOR as assessed will be presented.
Incidence of anti-drug antibodies (ADAs) against Gocatamig | At designated time points up to ~4 years
  Blood samples collected at designated timepoints will be used to determine the ADA response to gocatamig. The incidence of ADAs for gocatamig will be presented.
Incidence of ADAs against atezolizumab (for combination-treatment patients) | At designated time points up to ~4 years
  Blood samples collected at designated timepoints will be used to determine the ADA response to atezolizumab. The incidence of ADAs for atezolizumab will be presented.
Incidence of ADAs against I-DXd (for combination-treatment patients) | At designated time points up to ~4 years
  Blood samples collected at designated timepoints will be used to determine the ADA response to I-DXd. The incidence of ADAs for I-DXd will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (11):
- United States (11):
  - Cedar-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence, Portland, Oregon
  - Tennessee Oncology, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com